CLINICAL TRIAL: NCT05523050
Title: Effect of Active Surgical Intervention on Disease Remission in Patients With Crohn's Disease: A Single-Arm Trial
Brief Title: Active Surgical Intervention on Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WXSW-CD-001
Record Dates: First submitted 2022-08-25; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- active enterostomy (Other): active enterostomy before serious complications
  Interventions: Procedure: active surgical intervention

INTERVENTIONS:
Procedure: active surgical intervention — two kinds: one is colostomy, and the other one is colonic exclusion

SUMMARY:
The study is to determine whether active surgical intervention promotes disease remission in patients with Crohn's Disease (CD).The management of CD involves both maintenance medication and medication used to control flares of the disease. The goal of maintenance therapy in CD is to maintain steroid- free remission, clinically and endoscopically. This requires regular clinical assessment including history, physical examination and at times colonoscopic examination. Other tools of assessment include blood (e.g. CRP, WCC) and stool (calprotectin) testing for inflammatory markers and imaging including MRI, CT or ultrasound.

The choice of maintenance treatment in CD is determined by disease extent, disease course (frequency of flares), failure of previous maintenance treatment, severity of the most recent flare, treatment used for inducing remission during the most recent flare, safety of maintenance treatment, and cancer prevention. The mainstay of maintenance medication are the 5-aminosalicylic acid compounds (5-ASA) such as mesalazine or sulphasalazine.

These compounds are commonly taken orally in formulations that predominantly deliver the active 5-ASA component to the colon. Alternatively, or in addition, mesalazine preparations can be delivered topically via enema or suppository if the disease only involves the left side of the colon (although it is only PBS funded for topical therapy during a flare and not for maintenance of remission - even though it also works in this setting). The majority of patients can be managed with maintenance 5-ASA compounds most of the time. For patients who have repeated flares of disease on 5-ASA maintenance therapy (1 or more flares in a year needing steroids), thiopurine medication such as azathioprine or 6-mercapropurine should be used. These medications induce systemic immunosuppression, reduce the incidence and severity of flares of colitis but also slightly increase the risk of some infections and malignancy. Anti TNF agents such as infliximab or adalimumab have been shown to have benefit in maintaining remission in CD (and are licensed for this indication by the TGA), however these agents are very expensive and not funded by the pharmaceutical benefits scheme in Australia and so, are not readily available. The anti TNF agents also give an increased risk of infection, particularly latent TB reactivation.

Mild flares of CD can be managed with higher doses of oral 5-ASA compounds or the addition of topical 5-ASAs given via enema or suppository. More severe flares are usually managed with a course of systemic corticosteroid. These can be given intravenously in acute, severe disease or orally in less severe flares. The steroids should then be tapered over time and discontinued. There is no indication for long term steroid use in CD and prolonged steroid use is associated with a number of complications including infection, osteoporosis, obesity, diabetes, poor wound healing, thinning skin, mood changes and insomnia. Severe flares of CD not responsive to steroids may respond to rescue therapy with the addition of either cyclosporin or anti-TNF therapy.

Patients in whom colonic inflammation cannot be controlled adequately frequently undergo total colectomy. This may be done electively (for refractory disease) or emergently in acute fulminant colitis. Colectomy entails surgical risk that is higher in the emergent setting; this risk includes infection, wound breakdown and a mortality rate. Colectomy is considered "curative" for CD especially if they have an ileostomy stoma created, however, it frequently also leads to complications both short- and long-term. In addition, in patients in whom an ileal-anal pouch is fashioned up to 50% will subsequently develop pouchitis at 4 years post surgery.

Patient eligibility was determined during a 5-week screening period, during which time details on patient demographics, medical history, and previous and concomitant medications were obtained,and the following assessments were completed: viral serology, stool culture, Crohn's Disease Activity Index (CDAI) patient diary and clinical score, Simple Endoscopic Score for Crohn's Disease (SES-CD), colonoscopy and colonic biopsy, stool collection for faecal biomarkers, vital signs, and laboratory evaluations.

All participants need to be subjected to rigorous assessments mentioned above at week 4, week 8 and week 12 after receiving active surgical intervention (two kinds: one is colostomy, and the other one is colonic exclusion).

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe active CD (CDAI ≥ 150)
2. Endoscopic subscore meet the criteria (SES-CD ≥ 4)
3. Patients aged 18 to 75 years with established diagnosis of CD

Exclusion Criteria:

1. Mild active CD (CDAI < 150)
2. More than 25mg of prednisolone per day (or equivalent steroid)
3. Previous colonic surgery
4. Active gastrointestinal infection
5. Pregnancy
6. Anticoagulant therapy or duel antiplatelet therapy (i.e. aspirin and clopidogrel)
7. Current use of antibiotics
8. Anti-TNF therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-16 (Estimated); Primary Completion 2024-03-16 (Estimated); Study Completion 2024-05-16 (Estimated)

PRIMARY OUTCOMES:
SES-CD | 12 weeks
  Simple Endoscopic Score for Crohn's Disease

SECONDARY OUTCOMES:
CDAI | 12 weeks
  Crohn's Disease Activity Index

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, PhD, MD, Study Chair — The Affiliated Wuxi People's Hospital of Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No
To determine whether active surgical intervention promotes disease remission in patients with Crohn's Disease (CD).